CLINICAL TRIAL: NCT04592874
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of AL002 in Participants With Early Alzheimer's Disease
Brief Title: A Phase 2 Study to Evaluate Efficacy and Safety of AL002 in Participants With Early Alzheimer's Disease
Acronym: INVOKE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL002-2
Record Dates: First submitted 2020-09-17; First posted 2020-10-19 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AL002 Dose 1 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002
- AL002 Dose 2 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002
- AL002 Dose 3 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002
- Placebo (Placebo Comparator): Placebo every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL002 — Administered via intravenous (IV) infusion
  Arms: AL002 Dose 1; AL002 Dose 2; AL002 Dose 3
Drug: Placebo — Administered via intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
A phase 2 randomized, double blind, placebo controlled study evaluating the efficacy and safety of AL002 in participants with Early Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a phase 2 randomized, double blind, placebo controlled study evaluating the efficacy and safety of AL002 administered intravenously in participants with Early Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Early AD including evidence of brain amyloidosis by CSF or PET
* MMSE score ≥ 20 points, CDR Global Score of 0.5 - 1.0, and RBANS score on the DMI ≤95.
* Study partner who consents to study participation and who cares for/visits the participant at least 10 hours a week
* Written informed consent must be obtained and documented (from the participant or, where jurisdictions allow it, from their legal decision maker).

Exclusion Criteria:

* Dementia due to a condition other than AD including, but not limited to, FTD, Parkinson's disease, dementia with Lewy bodies, Huntington disease, or vascular dementia.
* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Current uncontrolled hypertension, diabetes mellitus or thyroid disease. Clinically significant heart disease, liver disease or kidney disease.
* History or evidence of clinically significant brain disease other than AD.
* Females who are pregnant or breastfeeding, or planning to conceive within the study period.
* Any experimental vaccine or gene therapy.
* History of unresolved cancer.
* Current use of anticoagulant medications.
* Residence in a skilled nursing facility, convalescent home, or long term care facility at screening; or requires continuous nursing care.
* Participant is positive for presence of APOE e4/e4 genotype.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Mummery, Principal Investigator
Locations (87):
- United States (29):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Woodlands Research Network, LLC - ERG, Rogers, Arkansas
  - ATP Clinical Research, Costa Mesa, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - South Florida Neurology Associates, Boca Raton, Florida
  - Brain Matters Research - ERG, Delray Beach, Florida
  - Charter Research, Lady Lake, Florida
  - ClinCloud, LLC, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - K2 Winter Garden Ocoee, Ocoee, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Axiom Clinical Research FL, Tampa, Florida
  - K2 The Villages, The Villages, Florida
  - Alzheimers Research and Treatment Center, Wellington, Florida
  - Conquest Clinical Research (Winter Park), Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - AMITA Health Clinical Research Institute, Elk Grove Village, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Boston Center for Memory, Newton, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Advanced Clinical Institute, Neptune City, New Jersey
  - Feinstein Institute For MR, Manhasset, New York
  - Columbia University College of Physicians and Surgeons, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - University of Cincinnati MC, Cincinnati, Ohio
  - Summit Research Network, Portland, Oregon
  - Abington Neurologic Associates, Abington, Pennsylvania
  - Clinical Trial Network, Houston, Texas
- Argentina (2):
  - Instituto Kremer, Córdoba
  - Centro de Psiquiatría Biológica Instituto Senecta, Mendoza
- Australia (4):
  - KaRa Institute of Neurological Disease, Macquarie Park, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Parkville, Victoria
  - SMarT Minds WA, Nedlands, Western Australia
- Canada (8):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - True North Clinical Research - Halifax, Halifax, Nova Scotia
  - True North Clinical Research - New Minas, New Minas, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Bruyère Research Institute, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Clinic, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
- France (5):
  - Hôpital Roger Salengro, Lille, Nord
  - Hopital Lariboisiere, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Gerontopole, Toulouse
- Germany (6):
  - Charité - Universitätsmedizin Berlin (CBF), Berlin
  - Charite Campus Buch, Berlin
  - University Clinic Heidelberg, Mannheim
  - LMU Klinikum der Universität München, München
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, München
  - Universitätsklinikum Ulm, Ulm
- Italy (10):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Azienda Policlinico Umberto I, Rome, Lazio
  - Ospedale S Giovanni Calibita Fatebenefratelli, Rome, Lazio
  - IRCCS - Centro S. Giovanni di Dio Fatebenefratelli, Brescia, Lombardy
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan
  - Ospedale Civile di Baggiovara, Modena
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale degli Infermi, Ponderano
- Netherlands (2):
  - Brain Research Center Den Bosch, 's-Hertogenbosch, North Brabant
  - Brain Research Center Amsterdam, Amsterdam
- CGM Research Trust, Christchurch, New Zealand
- Poland (4):
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne NeuroProtect, Warsaw, Masovian Voivodeship
  - EUROMEDIS Sp. z o.o., Szczecin, West Pomeranian Voivodeship
  - SOMED CR, Warsaw
- Spain (9):
  - Centro de Atencion Especializada Oroitu, Getxo, Basque Country
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Catalonia
  - Fundacion CITA Alzheimer Fundazioa, Donostia / San Sebastian, Guipuzcoa
  - Fundacion ACE Instituto Catalan de Neurociencias, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (7):
  - Re: Cognition Health - Guildford, Guildford, Surrey
  - Re:Cognition Health Bristol, Bristol
  - Re:Cognition Health London, London
  - The National Hospital for Neurology and Neurosurgery, London
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester
  - Glasgow Memory Clinic, Motherwell
  - Re:Cognition Health Plymouth, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shao Q, Chen S, Zheng Y, Xu W, Chen J, Shao W, Wang Q, Li C, Wang X. Crucial role of microglia-mediated myelin sheath damage in vascular dementia: Antecedents and consequences. Neural Regen Res. 2026 Mar 1;21(3):1000-1012. doi: 10.4103/NRR.NRR-D-24-01109. Epub 2025 Mar 25. PMID 40145953
- [Derived] Brodtmann A, Darby D, Oboudiyat C, Mahoney CJ, Le Heron C, Panegyres PK, Brew B. Assessing preparedness for Alzheimer disease-modifying therapies in Australasian health care systems. Med J Aust. 2023 Apr 3;218(6):247-249. doi: 10.5694/mja2.51880. Epub 2023 Mar 19. No abstract available. PMID 36934371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 328 participants were planned to be enrolled: Part 1: Approximately 40 participants were to be randomized in a 1:1:1:1 ratio to receive either 15 mg/kg AL002, 40 mg/kg AL002, 60 mg/kg AL002, or placebo. Part 2: Approximately 288 participants were to be enrolled with the same allocation ratio (1:1:1:1) used in Part 1.
Pre-assignment Details: Screening period of up to 8 weeks prior to the optional Predose Baseline Visit or to Day 1 visit.
Groups:
- AL002 Dose 1: 15 mg/kg; AL002 Dose 2: 40 mg/kg; AL002 Dose 3: 60 mg/kg: AL002 every 4 weeks
Period: Overall Study
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Started | 97 | 94 | 77 | 88
Completed | 51 | 53 | 50 | 72
Not Completed | 46 | 41 | 27 | 16

BASELINE CHARACTERISTICS:
Population: This field outlines the number of participants that were treated in each arm
Groups:
- Total: Total of all reporting groups
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo | Total
Number analyzed (Participants) | 97 | 94 | 77 | 88 | 356
Age, Categorical [Count of Participants; unit: Participants] — This field outlines the age categories of the participants per arm Population: This field outlines the age categories of the participants per arm
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 24 | 24 | 15 | 15 | 78
    >=65 years | 73 | 70 | 62 | 73 | 278
Sex: Female, Male [Count of Participants; unit: Participants] — This field outlines the sex of the participants per arm Population: This field outlines the sex of the participants per arm
  Participants
    Female | 45 | 52 | 39 | 44 | 180
    Male | 52 | 42 | 38 | 44 | 176
Race (NIH/OMB) [Count of Participants; unit: Participants] — This field outlines the race of the participants per arm Population: This field outlines the race of the participants per arm
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 3 | 0 | 0 | 0 | 3
    White | 88 | 92 | 72 | 82 | 334
    More than one race | 0 | 0 | 0 | 1 | 1
    Unknown or Not Reported | 6 | 2 | 3 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This is the ethnicity of the participants per arm Population: This is the ethnicity of the participants per arm
  Participants
    Hispanic or Latino | 4 | 5 | 4 | 4 | 17
    Not Hispanic or Latino | 87 | 86 | 70 | 81 | 324
    Unknown or Not Reported | 6 | 3 | 3 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Measured by the Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score
Description: Change from baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) score at Weeks 24, 48, 72 and 96.
  The CDR-SB is a tool used to measure disease severity in Alzheimer's disease. This scale assesses three domains of cognition and three domains of function. The domains are rated on a 5 point scale in which the higher the score corresponds to greater cognitive impairment. The scale range is from 0 to 18 where 0 is considered normal and 18 indicates severe dementia.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 66 | 73 | 68 | 83
  Week 24 Change from Baseline | 1.02 (0.197) | 0.80 (0.190) | 1.07 (0.196) | 1.15 (0.180)
  Week 48 Change from Baseline: number analyzed (Participants) | 62 | 60 | 59 | 73
  Week 48 Change from Baseline | 1.68 (0.256) | 1.61 (0.256) | 1.95 (0.259) | 1.68 (0.236)
  Week 72 Change from Baseline: number analyzed (Participants) | 32 | 34 | 31 | 42
  Week 72 Change from Baseline | 2.61 (0.366) | 2.93 (0.358) | 2.12 (0.372) | 2.25 (0.324)
  Week 96 Change from Baseline: number analyzed (Participants) | 20 | 18 | 18 | 26
  Week 96 Change from Baseline | 3.17 (0.488) | 3.61 (0.498) | 3.31 (0.506) | 3.48 (0.435)
Statistical Analysis 1: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7975, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-1.49 to 1.15]
Statistical Analysis 2: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.6341, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.61 to 0.98]
Statistical Analysis 3: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.8489, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-1.18 to 1.43]

2. Secondary Outcome: Change in Mini-Mental Status Examination (MMSE) Score
Description: Change from baseline in Mini-Mental Status Examination (MMSE) score at Weeks 24, 48, 72, and 96
  The MMSE is a test that assesses orientation, registration, attention and calculation, recent memory, language and constructional praxis. There is a total possible score of 30 with a lower score correlating to a higher cognitive impairment. A score of 24 to 30 is considered normal or no cognitive impairment. A score of 18 to 24 indicates mild impairment. A score of 0 to 17 indicates a severe impairment.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 67 | 74 | 69 | 83
  Week 24 Change from Baseline | -2.70 (0.396) | -3.03 (0.381) | -2.78 (0.393) | -2.65 (0.364)
  Week 48 Change from Baseline: number analyzed (Participants) | 63 | 62 | 59 | 74
  Week 48 Change from Baseline | -4.06 (0.541) | -3.91 (0.535) | -3.74 (0.549) | -3.33 (0.501)
  Week 72 Change from Baseline: number analyzed (Participants) | 32 | 34 | 31 | 42
  Week 72 Change from Baseline | -5.15 (0.772) | -5.47 (0.751) | -4.99 (0.780) | -4.89 (0.692)
  Week 96 Change from Baseline: number analyzed (Participants) | 20 | 18 | 18 | 26
  Week 96 Change from Baseline | -5.88 (0.906) | -7.22 (0.914) | -5.81 (0.932) | -5.47 (0.814)
Statistical Analysis 1: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7417, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-2.81 to 2.01]
Statistical Analysis 2: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.1559, Mixed Models Analysis; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-4.16 to 0.67]
Statistical Analysis 3: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7850, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-2.78 to 2.11]

3. Secondary Outcome: Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Score
Description: Change from baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score at Weeks 24, 48, 72 and 96
  The RBANS test is a collection of 12 subsets representing 5 neurological domains: immediate memory, visuospatial/constructional, language, attention, and delayed memory. The scores are converted to a scale that can range from 40 to 160. The lower the score the greater the cognitive impairment.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 62 | 70 | 60 | 78
  Week 24 Change from Baseline | -3.37 (0.857) | -2.34 (0.820) | -2.65 (0.870) | -3.05 (0.782)
  Week 48 Change from Baseline: number analyzed (Participants) | 53 | 55 | 50 | 69
  Week 48 Change from Baseline | -7.15 (0.939) | -6.13 (0.921) | -5.78 (0.957) | -5.05 (0.844)
  Week 72 Change from Baseline: number analyzed (Participants) | 25 | 28 | 24 | 36
  Week 72 Change from Baseline | -6.46 (1.339) | -6.56 (1.281) | -5.94 (1.357) | -5.86 (1.149)
  Week 96 Change from Baseline: number analyzed (Participants) | 15 | 13 | 15 | 23
  Week 96 Change from Baseline | -8.12 (1.915) | -7.23 (2.011) | -6.56 (1.936) | -7.47 (1.574)
Statistical Analysis 1: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7934, Mixed Models Analysis; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-5.58 to 4.28]
Statistical Analysis 2: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.9259, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-4.84 to 5.32]
Statistical Analysis 3: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7147, Mixed Models Analysis; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-4.04 to 5.87]

4. Secondary Outcome: Change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) Score
Description: Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) score at Weeks 24, 48, 72, and 96
  The ADAS-Cog13 is a scale that includes 13 items to assess cognitive function. These domains include memory, language, praxis, and orientation, as well as a number cancellation task and a delayed free recall task. There is a total score range of 0 to 85. A higher score on this scale indicates greater cognitive impairment. There are currently no universally accepted severity bands for ADAS-Cog13 as it is used to track changes in disease and not for severity.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 68 | 71 | 67 | 81
  Week 24 Change from Baseline | 1.09 (0.710) | 3.04 (0.697) | 3.54 (0.717) | 1.93 (0.659)
  Week 48 Change from Baseline: number analyzed (Participants) | 60 | 61 | 59 | 73
  Week 48 Change from Baseline | 3.86 (0.960) | 6.06 (0.950) | 5.67 (0.967) | 3.79 (0.880)
  Week 72 Change from Baseline: number analyzed (Participants) | 30 | 33 | 31 | 37
  Week 72 Change from Baseline | 7.31 (1.325) | 8.30 (1.285) | 7.34 (1.321) | 6.26 (1.205)
  Week 96 Change from Baseline: number analyzed (Participants) | 19 | 18 | 18 | 24
  Week 96 Change from Baseline | 9.59 (1.543) | 10.02 (1.541) | 11.55 (1.563) | 8.62 (1.397)
Statistical Analysis 1: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.6403, Mixed Models Analysis; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-3.14 to 5.09]
Statistical Analysis 2: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.5016, Mixed Models Analysis; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-2.71 to 5.51]
Statistical Analysis 3: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.1631, Mixed Models Analysis; Mean Difference (Final Values) = 2.94, 95% CI 2-sided [-1.21 to 7.08]

5. Secondary Outcome: Change in Alzheimer's Disease Cooperative Study - Activities of Daily Living - Mild Cognitive Impairment (ADCS-ADL-MCI) Score
Description: Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living - Mild Cognitive Impairment (ADCS-ADL-MCI) score at Weeks 24, 48, 72, and 96
  The ADCS-ADL-MCI is a scale for participants with mild cognitive impairment that observes their performance in completing activities associated with daily living. This scale is a multiple choice questionnaire and has a range of 0 to 53. A lower score on this scale indicates greater cognitive impairment.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 66 | 70 | 67 | 81
  Week 24 Change from Baseline | -1.60 (0.608) | -0.99 (0.594) | -2.45 (0.607) | -0.67 (0.559)
  Week 48 Change from Baseline: number analyzed (Participants) | 62 | 61 | 58 | 74
  Week 48 Change from Baseline | -2.95 (0.808) | -3.11 (0.811) | -3.46 (0.828) | -2.73 (0.744)
  Week 72 Change from Baseline: number analyzed (Participants) | 32 | 34 | 31 | 41
  Week 72 Change from Baseline | -6.41 (1.183) | -6.57 (1.159) | -6.80 (1.201) | -5.36 (1.063)
  Week 96 Change from Baseline: number analyzed (Participants) | 20 | 18 | 18 | 25
  Week 96 Change from Baseline | -8.50 (1.517) | -7.80 (1.549) | -7.44 (1.570) | -7.97 (1.368)
Statistical Analysis 1: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7945, Mixed Models Analysis; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-4.57 to 3.51]
Statistical Analysis 2: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.9371, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-3.92 to 4.25]
Statistical Analysis 3: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.7991, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-3.58 to 4.64]

6. Secondary Outcome: Change in Alzheimer's Disease Composite Score (ADCOMS) Score
Description: Change from baseline in Alzheimer's Disease Composite Score (ADCOMS) score at Weeks 24, 48, 72, and 96
  The ADCOMS scale is a composite score of 12 components that include 4 items from the ADAS-Cog13, 2 items from the MMSE, and all 6 items from the CDR-SB scales. The range of the ADCOMS is between 0 and 1.97. The higher the score the greater the cognitive impairment.
Time Frame: Study completion up to 96 weeks
Population: Adult participants with early Alzheimer's Disease excluding apolipoprotein E homozygotes
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
Number analyzed (Participants) | 89 | 87 | 92 | 88
Score on a scale
  Week 24 Change from Baseline: number analyzed (Participants) | 66 | 70 | 67 | 81
  Week 24 Change from Baseline | 0.11 (0.020) | 0.11 (0.019) | 0.14 (0.020) | 0.13 (0.018)
  Week 48 Change from Baseline: number analyzed (Participants) | 58 | 59 | 59 | 72
  Week 48 Change from Baseline | 0.19 (0.027) | 0.20 (0.027) | 0.25 (0.027) | 0.20 (0.024)
  Week 72 Change from Baseline: number analyzed (Participants) | 27 | 32 | 30 | 37
  Week 72 Change from Baseline | 0.25 (0.041) | 0.36 (0.039) | 0.25 (0.040) | 0.26 (0.036)
  Week 96 Change from Baseline: number analyzed (Participants) | 19 | 18 | 18 | 24
  Week 96 Change from Baseline | 0.32 (0.052) | 0.43 (0.052) | 0.39 (0.053) | 0.35 (0.047)
Statistical Analysis 1: Comparison: AL002 Dose 1: 15 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.6458, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.17 to 0.11]
Statistical Analysis 2: Comparison: AL002 Dose 2: 40 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.2779, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.06 to 0.21]
Statistical Analysis 3: Comparison: AL002 Dose 3: 60 mg/kg vs Placebo; This is using the Week 96 timepoint; Test type: Superiority; p = 0.5355, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.10 to 0.18]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) have been reported from the screening period up to 8 weeks prior to dosing through 8 weeks after the last dose administration which could be up to 115 weeks of study participation.
Arm/Group | AL002 Dose 1: 15 mg/kg | AL002 Dose 2: 40 mg/kg | AL002 Dose 3: 60 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/97 | 1/94 | 1/77 | 1/88
Serious Adverse Events (participants affected / at risk) | 14/97 | 12/94 | 10/77 | 7/88
Other Adverse Events (participants affected / at risk) | 66/97 | 75/94 | 59/77 | 64/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL002 Dose 1: 15 mg/kg (N=97) | AL002 Dose 2: 40 mg/kg (N=94) | AL002 Dose 3: 60 mg/kg (N=77) | Placebo (N=88)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Amyloid related imaging abnormality - edema/effusion (Nervous system disorders) | 1 | 1 | 0 | 0
Amyloid related imaging abnormality - microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Colonic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AL002 Dose 1: 15 mg/kg (N=97) | AL002 Dose 2: 40 mg/kg (N=94) | AL002 Dose 3: 60 mg/kg (N=77) | Placebo (N=88)
Fall (Injury, poisoning and procedural complications) | 5 | 19 | 7 | 11
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 9 | 10 | 2
Hypertension (Vascular disorders) | 4 | 6 | 7 | 6
Amyloid related imaging abnormality-microhaemorrages and haemosiderin deposits (Nervous system disorders) | 28 | 28 | 21 | 4
Amyloid related imaging abnormality-edema/effusion (Nervous system disorders) | 21 | 22 | 17 | 1
Headache (Nervous system disorders) | 10 | 13 | 4 | 10
Dizziness (Nervous system disorders) | 6 | 7 | 6 | 7
Syncope (Nervous system disorders) | 1 | 2 | 1 | 6
Fatigue (General disorders) | 3 | 4 | 4 | 4
Cataract (Eye disorders) | 7 | 6 | 7 | 3
Vomiting (Gastrointestinal disorders) | 6 | 8 | 7 | 1
Nausea (Gastrointestinal disorders) | 5 | 6 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 1 | 7
Confusional state (Psychiatric disorders) | 1 | 3 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 6
Covid-19 (Infections and infestations) | 11 | 12 | 13 | 19
Nasopharyngitis (Infections and infestations) | 6 | 2 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 5 | 7
Urinary tract infection (Infections and infestations) | 5 | 4 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alector's agreements with principal investigators may vary but will not prohibit any investigator from publishing. Alector supports the publication of the results from all centers in a multi-center trial, and its agreements include provisions to enable the multi-center publication to occur before publication of data from a single site.

DOCUMENTS (2):
  • Study Protocol (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04592874/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04592874/SAP_001.pdf